CLINICAL TRIAL: NCT03721003
Title: Intracranial Pressure Monitoring in Sever Traumatic Brain Injury Single Centre Experience
Brief Title: Intracranial Pressure Monitoring in Sever Traumatic Brain Injury Single Center Experience
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mosab Samir, doctor, Assiut University
Other Study IDs: IPMISTBISCE
Record Dates: First submitted 2018-09-29; First posted 2018-10-26 (Actual); Last update posted 2018-10-26 (Actual); Status verified 2018-10

CONDITIONS: Head Injury Trauma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: ICP monitoring — 4- Use the Touhy needle to tunnel under the scalp from the Burr Hole site to the desired MICROSENSOR exit site.
  5- Place the tip of the MICROSENSOR in the Parenchyma through the puncture in the Dura

SUMMARY:
Intracranial pressure (ICP) is defined as the pressure inside the skull, and therefore, the pressure inside the brain tissue and the cerebrospinal fluid (CSF). The relationship between CSF and intracranial blood volumes is described by the Monroe Kellie doctrine; because the brain is incompressible, when the skull is intact, the sum of the volumes of brain, CSF, and intracranial blood is constant.

DETAILED DESCRIPTION:
ICP >15 mmHg is considered to be elevated, and this is considered an important cause of secondary injury leading to irreversible brain injury and death. ICP monitoring is used in a number of conditions; traumatic brain injury, intracerebral haemorrhage, subarachnoid haemorrhage, hydrocephalus, malignant infarction, cerebral oedema, CNS infections, hepatic encephalopathy, to name a few, and in all of these conditions ICP monitoring in the light of other parameters can influence management for better outcomes.

There are 4 ways to monitor intracranial pressure:

1. An intra-parenchymal method, the catheter is placed into the brain parenchyma through a burr hole; it has a lower complication rate, lower infection rate, and no chance of catheter occlusion or leakage. Neurological injury is minimized because of the small diameter of the probe. In addition, malposition of the transducer has less impact on errors of measurement.
2. An intra-ventricular method, the catheter is placed into one of the ventricles (lat. Ventricle). The catheter can also be used for therapeutic CSF drainage and for administration of drugs.
3. Subdural method, this method is used if monitoring needs to be done right away. A hollow screw is inserted through a burr hole and placed through the Dura mater.
4. An epidural sensor is inserted between the skull and dural tissue. This procedure is less invasive than other methods.

ICP monitoring methods is associated with a number of complications. These include risk of infection, haemorrhage, obstruction, difficulty in placement, malposition, etc.

The use of an ICP monitor is associated with significantly lower mortality when compared with patients treated without an ICP monitor

ELIGIBILITY:
Inclusion Criteria:

1. Age >18
2. GCS < 8
3. patient with severe brain insult ( Marshall class II to IV)
4. patients admitted within 24 hours from the trauma time

Exclusion Criteria:

1. Patients admitted for surgery (ex; surgical EDH) .
2. patient diagnosed as brain death

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: history of present illness will be taken clinical assesment will be done ct brain will be done after that ICP monitor will be applied
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2020-01-01 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
analyse role of ICP monitoring of patient with diffuse traumatic brain injury | one year
  study the significance of application of ICP monitor on outcome of patients with diffuse traumatic brain injury using glascow coma scale The Glasgow Coma Scale (GCS) is a neurological scale which aims to give a reliable and objective way of recording the conscious state of a person for initial as well as subsequent assessment. A patient is assessed against the criteria of the scale, and the resulting points give a patient score between 3 (indicating deep unconsciousness) and either 14 (original scale) or 15 (more widely used modified or revised scale)

IPD SHARING:
Plan to Share IPD: No